CLINICAL TRIAL: NCT01694641
Title: Time Lapse Embryo Monitoring Versus Standard Embryo Monitoring for Selection for Single Blastocyst Transfer
Brief Title: Embryo Selection by Time Lapse Monitoring for Single Embryo Transfer ("SET")
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A general TL algorithm with higher predicting power became available in 2015 (Petersen et al.) and speed of recruitment was slower than expected.
Sponsor: Dunamenti REK Istenhegyi IVF Center (Other)
Collaborators: Forgacs Intezet Kft. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TL-SET
Record Dates: First submitted 2012-09-21; First posted 2012-09-27 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Clinical Pregnancy After Single Embryo Transfer
Keywords: time lapse monitoring; blastocyst; single embryo transfer; clinical pregnancy; implantation rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- time-lapse morphokinetic evaluation (Experimental): Embryo selection for transfer based on a combind score made up of scores for kinetic parameters and standard morphology as seen on time-lapse: upon fertilization embryos in a petri dish that allows individual assessment (Primo Vision Dish) are placed onto an automated time-lapse equipment in an incubator. The time-lapse equipment performs imaging in 10 minutes intervals. The software is presenting the up-to-date images and allows the operator to assess the "time-lapse" movie of the developmental history of the embryos to perform annotations and apply evaluation/selection algorithm. This morpho-kinetic TL algorithm (made up of standard moprhology as seen on time lapse and kinetci scores) is used for embryo selection, which actually describes the intervention.
  Interventions: Other: time-lapse morphokinetic evaluation
- standard embryo monitoring (No Intervention): Upon fertilization embryos are observed once on days 1-3-5 by the embryologist to check for development. The single embryo for transfer is selected based on actual morphology as seen under light microscope.

INTERVENTIONS:
Other: time-lapse morphokinetic evaluation — embryo selection for transfer based on a combind score made up of scores for kinetic parameters and standard morphology as seen on time-lapse
  Other Names: time-lapse morphokintic score
  Arms: time-lapse morphokinetic evaluation

SUMMARY:
A multiple pregnancy is an undesired outcome of assisted reproduction. Current embryo selection technologies are inefficient in identifying the embryo with the highest implantation potential. Time lapse (TL) embryo monitoring provides additional information about embryo development and therefore may aid embryo selection. The investigators aim is to study whether TL monitoring is superior to traditional embryo observation when a single blastocyst is selected for transfer (ET).

DETAILED DESCRIPTION:
Prospective RCT comparing two embryo selection methods (TL algorithm vs standard morphology based) for SET. Infertile couples scheduled to undergo IVF or intracytoplasmic sperm injection (ICSI) and met the inclusion-exclusion criteria were enrolled. Randomization to Groups 1 or 2 was performed prior to the start of stimulation. Randomization was carried out in blocks of two, by selecting TL or control assignments from closed, opaque envelopes. Patients were blinded to allocation. Standard luteal long (Suprefact, Sanofi Aventis) and flexible gonadotropin-releasing hormone (GnRH) antagonist (Cetrotide, Merck Serono) protocols and recombinant FSH(Gonal-f, Merck Serono) were used for stimulation. Embryos were placed into individual wells of a 9-well Primo Vision culture dish (Vitrolife AB, Sweden) on day 1 of culture, after checking for fertilization. Out of incubator handling was same in the groups;: day 1: fertilization check; day 3: culture medium change; day 5: transfer. On days 3 and 5, the embryos were morphologically assessed under an inverted microscope. Embryos in TL group were imaged at 10-minute intervals. The Primo Vision software was used for the analysis of TL images. The first appearance of the 2, 3, 4 and 5 cell stages (t2, t3, t4 and t5, respectively) were annotated. Timing of the kinetic events was calculated from the time of the fertilization (t0). (for TL parameter definitions see supplement) There were no adjustments of the kinetic events depending on the method of fertilization. Blastocyst morphology was assessed using the Gardner score. Fragmentation was assessed when it reached the highest grade in the sequence of the TL images. Cytoplasmic abnormalities (vacuoles) were also recorded. The TL reference ranges were defined and fixed before the start of the recruitment, Embryos in the control group were selected based on actual morphology. The primary end point was pregnancy rate (PR; rise in β human chorionic gonadotropin [hCG]) per patient based on intention to treat. Further endpoints were ongoing pregnancy rate (OPR; pregnancy that progresses beyond 12 weeks gestation), pregnancy loss (loss of pregnancy after an initial rise in βhCG up to 12 weeks gestation), live birth rate (LBR), gestational age (GA) at delivery and birth weight of the offspring.

When calculating sample size we assumed a 13% increase in pregnancy rate from an expected 42% to 55%. We planned to run the study with 1:1 ratio between the groups and do one interim monitoring with 0.1 information fraction. Using two-sided test and Pocock boundaries for estimation, 282 patients in each group was calculated (power of 80%, p of 5%). Assuming a 10% dropout rate we needed to enroll 620 patients.

Based on the results of the interim monitoring (61 cases in two arms) the pregnancy rate in the TL group was 15% higher than in controls (58.3% vs. 44.0%). Assuming 58% pregnancy rate in the TL group and 44% in controls, a sample size of 210 per group, was needed to achieve a power of 80%, at a significance level of 5%. Assuming 10% dropout rate a total sample of size of 462 patients were needed.

The groups were compared based on maximum likelihood estimation principles. We hypothesized and then showed that the patients in the treatment arms were similar at baseline, on average, with respect to variables that might influence outcome. Chi-square tests, likelihood-ratio tests and exact tests were used for the analysis of categorical variables. Continuous variables were compared using independent group t-test and. analysis of variance. Normality and homogeneity of variances were examined.

At the interim analysis of the trial the primary endpoint (pregnancy rate) between TL and control group was compared with Fisher's exact test. After closing the trial the primary endpoint (pregnancy rate) among the groups was compared with Fisher's exact test. Bonferroni correction was used for the p-value at the end of the trial. All other p-values were considered exploratory in nature. During the analyses the extent and distribution of missing data were also examined. No imputations were made for missing data.

ELIGIBILITY:
Inclusion Criteria:

* Age < 36 yrs
* baseline FSH <10 IU/l
* regular 25-35 day cycles
* less than 2 previous failed IVF cycles
* intact uterus
* an indication for IVF
* BMI <18- <30 kg/m2
* acceptance of single embryo transfer

Exclusion Criteria:

* PCOS
* Sperm obtained by surgical extraction
* chromosome abnormality
* Presence of hydrosalpinx
* stage III/IV endometriosis
* Less than 3 good quality day 3 embryos
* only one good quality day 5 embryos
* lack of consent

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kovacs, MD, Principal Investigator — Kaali Inst. IVF Center
Locations (2):
- Hungary (2):
  - Kaali Institute IVF Center, Budapest
  - Forgacs Intezet, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pribenszky C, Matyas S, Kovacs P, Losonczi E, Zadori J, Vajta G. Pregnancy achieved by transfer of a single blastocyst selected by time-lapse monitoring. Reprod Biomed Online. 2010 Oct;21(4):533-6. doi: 10.1016/j.rbmo.2010.04.015. Epub 2010 Apr 24. PMID 20638906
- [Background] Pribenszky C, Losonczi E, Molnar M, Lang Z, Matyas S, Rajczy K, Molnar K, Kovacs P, Nagy P, Conceicao J, Vajta G. Prediction of in-vitro developmental competence of early cleavage-stage mouse embryos with compact time-lapse equipment. Reprod Biomed Online. 2010 Mar;20(3):371-9. doi: 10.1016/j.rbmo.2009.12.007. Epub 2010 Jan 25. PMID 20089456
- [Background] Meseguer M, Herrero J, Tejera A, Hilligsoe KM, Ramsing NB, Remohi J. The use of morphokinetics as a predictor of embryo implantation. Hum Reprod. 2011 Oct;26(10):2658-71. doi: 10.1093/humrep/der256. Epub 2011 Aug 9. PMID 21828117

RESULTS

PARTICIPANT FLOW:
Groups:
- Time Lapse Embryo Observation: Embryo selection for transfer based on a combind score made up of scores for kinetic parameters and standard morphology as seen on time-lapse: upon fertilization embryos are placed in an incubator that is hooked up to a monitor that allows continuous embryo observation. A morpho-kinetic TL algorithm (made up of standard moprhology as seen on time lapse and kinetci scores) is used for embryo selection.
  time-lapse morphokinetic evaluation: embryo selection for transfer based on a combind score made up of scores for kinetic parameters and standard morphology as seen on time-lapse
Period: Overall Study
Arm/Group | Time Lapse Embryo Observation | Standard Embryo Monitoring
Started | 80 | 81
Completed | 68 | 71
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Population: 161 patients were randomized. Each patient participated only once in the RCT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Time Lapse Embryo Observation | Standard Embryo Monitoring | Total
Number analyzed (Participants) | 80 | 81 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 81 | 161
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (2.7) | 32.1 (2.5) | 31.7 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 81 | 161
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 80 | 81 | 161

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate
Description: rise in beta HCG 12-14 days after transfer
Time Frame: 12-14 days after transfer
Population: All patients randomized are analyszs (intention to treat analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | Time Lapse Embryo Observation | Standard Embryo Monitoring
Number analyzed (Participants) | 80 | 81
Participants | 34 | 26

2. Secondary Outcome: Live Birth
Description: live birth after 24 weeks gestation
Time Frame: delivery after 24 weeks
Population: All patients randomzed regardless whether completed the study or not according to their assignment (intention to treat population).
Measure: Count of Participants; unit: Participants
Arm/Group | Time-lapse Morphokinetic Evaluation | Standard Embryo Monitoring
Number analyzed (Participants) | 80 | 81
Participants | 34 | 26

3. Other Pre Specified Outcome: Time Lapse Score
Description: a score based on 8 observations by time lapse monitoring
Time Frame: the time lapse score is assessed on the day of embryo transfer (day 5 after the egg retrieval)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Perinatal Outcome
Description: gestational age at delivery, birth weight,
Time Frame: perinatal outcome assessed after delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Time Lapse Embryo Observation | Standard Embryo Monitoring
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/81
Other Adverse Events (participants affected / at risk) | 0/80 | 0/81

LIMITATIONS AND CAVEATS:
The downside of the study demographics is that we limited the study population to good prognosis cases therefore the conclusions can only be applied to similar patients. Stopped the study before meeting calculated sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes